CLINICAL TRIAL: NCT03230617
Title: Evaluation Of Dynamic Hyperinflation In Mechanically Ventilated Chronic Obstructive Pulmonary Disease Patients
Brief Title: Dynamic Hyperinflation In Mechanically Ventilated Chronic Obstructive Pulmonary Disease Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nisreen Mtk, principal investigator, Assiut University
Other Study IDs: EDHMVCP
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ventilators, Mechanical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intrinsic positive end expiratory pressure > 5: chronic obstructive pulmonary disease patient with intrinsic positive end expiratory pressure more than5
  Interventions: Device: Mechanical ventilator
- Auto positive end expiratory pressure < 5: chronic obstructive pulmonary disease patient with intrinsic positive end expiratory pressure less than5
  Interventions: Device: Mechanical ventilator

INTERVENTIONS:
Device: Mechanical ventilator — Mechanical ventilation, in the healthcare setting or home, helps patients breathe by assisting the inhalation of oxygen into the lungs and the exhalation of carbon dioxide. Depending on the patient's condition, mechanical ventilation can help support or completely control breathing.

SUMMARY:
Chronic obstructive pulmonary disease is a common respiratory condition that is characterized by inflammation of the large and small peripheral airways , the alveoli and adjacent capillary networks. Severe airflow obstruction that imposes a significant load on the respiratory system is a major manifestation of Chronic obstructive pulmonary disease. The reduced expiratory airflow also causes air trapping at the end of expiration , producing alveolar pressure that are higher than atmospheric pressure before the next breath. This condition is intrinsic positive end-expiratory pressure .

ELIGIBILITY:
Inclusion Criteria:

* patient with acute exacerbation of Chronic obstructive pulmonary disease and respiratory failure who are intubated and mechanically ventilated.

Exclusion Criteria:

* patient with neuromuscular diseases.
* patient with pulmonary vascular diseases e.g pulmonary embolism.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patient who diagnosed as chronic obstructive pulmonary disease admitted to the respiratory intensive care unit, chest department, Assiut university hospital, who are mechanically ventilated.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
The duration of mechanical ventilation | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Reddy VG. Auto-PEEP: how to detect and how to prevent--a review. Middle East J Anaesthesiol. 2005 Jun;18(2):293-312. PMID 16438005